CLINICAL TRIAL: NCT03675698
Title: Nasal Cavity Evaluation by CT Scan/ Magnetic Resonance Imaging to Access the Size of Nasotracheal Tube for Nasal Intubation
Brief Title: Radiological Images for Nasotracheal Tube Size Estimation
Acronym: RINSE
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Amit Kumar Mittal, Consultant in-charge, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RES/SCM/30/2018/82
Record Dates: First submitted 2018-09-15; First posted 2018-09-18 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Nasotracheal Tube Passage Through Nasal Cavity
Keywords: Nasotracheal tube size based on radiological images of nose.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nasotracheal Intubation — side of nostril and size of endotracheal tube estimation for nasotracheal intubation will be done based on radiological imaging ( CT/MRI head)
  Other Names: Malinckrodt flexometallic tube

SUMMARY:
This trial is planned to estimate the size of nasotracheal tube (NTT) by calculating the diameter of both nasal cavity in radiological images of nose (CT scan/MRI) at the level below the inferior turbinate and floor of nose in coronal planes. Smallest diameter will be considered to calculate the outer diameter of NTT, hence the size .

DETAILED DESCRIPTION:
The planned trial will estimate the size of nasotracheal tube (NTT) by calculating the diameter of both nasal cavity in radiological images of nose (CT scan/MRI) at the level below the inferior turbinate and floor of nose at different levels in coronal planes. Smallest diameter will be considered to calculate the outer diameter of NTT, hence the size. The side of nasotracheal intubation will be decided after view the radiological images and the estimated size of NTT will be used. Finally the ease of intubation and complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. patients requiring nasal intubation for oromaxillofacial surgeries

   Exclusion Criteria:
   * 1. Midface instability
2. Coagulopathy
3. Suspected basilar skull fractures
4. Large nasal polyps
5. Suspected nasal foreign bodies
6. Recent nasal surgery
7. History of frequent episodes of epistaxis
8. Prosthetic heart valves (increased risk of bacteremia during the insertion).
9. Patients with deranged liver and renal functions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: oncosurgical patients with oral malignancies who required nasotracheal intubation for COMMANDO surgeries.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Successful nasal intubation by selecting the correct size of nasotracheal tube estimated by measuring the diameter of nasal cavity in coronal section just below the inferior turbinate in radiological images. | After enrolment of the patient and before intubation
  The diameter of both nasal cavities in coronal section of CT/MRI will be calculated at the level just below the inferior turbinate in anterior nasal cavity when inferior turbinates just appeared in the radiological image, than at level of maxillary sinus and just before cohanal opening in radiological images. Minimal diameter will be used to estimate the size of nasotracheal tube before intubation.The images will also be used to select the side of nasal intubation after ruling out any nasal pathology like DNS, Spurs and marked turbinate hypretrophy.

SECONDARY OUTCOMES:
To find the complications associated with nasal intubations that were performed after assessing the radiological images. | At the time of intubation
  The radiological images will be studied prior to intubation, the appropriate size of the nasotracheal tube will be selected and after ruling out any nasal pathology like DNS , spurs, concha bullosa side of nasal intubation will be decided.

CONTACTS AND LOCATIONS:
Locations (1):
- Amit, Rohini, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans SW, McCahon RA. Management of the airway in maxillofacial surgery: part 2. Br J Oral Maxillofac Surg. 2018 Jul;56(6):469-474. doi: 10.1016/j.bjoms.2018.05.012. Epub 2018 Jun 12. PMID 29907468